CLINICAL TRIAL: NCT06165367
Title: Impact of Hyaluronan-enriched Medium on Pregnancy Outcomes Following Euploid Blastocyst Transfers
Brief Title: Hyaluronan-enriched Medium and Euploid Blastocyst Transfers
Acronym: GluePloid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Daniela Nogueira, Global Scientific Laboratory Director ART Fertility Clinics, ART Fertility Clinics LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART FERTILITY CLINICS
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Infertility; Implantation Rate; Clinical Pregnancy Rate; Live Birth Rate; Blastocysts; FET
Keywords: HRT; PGT-A; Next-generation sequencing (NGS); Miscarriage rate; single embryo transfer (SET); EmbryoGlue; BMI; Embryo quality; Hyaluronan-enriched medium; Transfer medium
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified according to the in-house embryo prognosis classification. Our internal data shows top quality embryos have 65% ongoing pregnancy rate and good quality embryos have 55% ongoing pregnancy rate. We assume a 20% relative increase over the baseline with the intervention which corresponds to 78% and 66% ongoing pregnancy rates for top and good quality euploid embryos, respectively. Total sample size requires in each group corresponds to 295 and 488 transfers of top and good quality embryos for a total of 783. Two interim analyses are planned when 35% (n=274) and 70% (n=548) of the target sample size is achieved to calculate conditional power. If conditional power is estimated to be lower than 15% at first interim analysis or lower than 30% in the second interim analysis, the trial will be stopped due to futility.
Who Masked: Participant, Care Provider
Masking Description: The study will be double-blinded (blinded to patient and doctor performing transfer).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blastocysts exposed to normal media (NEG) (No Intervention): Blastocysts exposed to routine-in use medium No intervention
- Blastocysts exposed to EmbryoGlue (EG) (Active Comparator): Blastocysts exposed to EmbryoGlue
  Interventions: Drug: EmbryoGlue Medium

INTERVENTIONS:
Drug: EmbryoGlue Medium — Embryos will be exposed to hyaluronic-enriched media (EmbryoGlue) before and during embryo transfer
  Arms: Blastocysts exposed to EmbryoGlue (EG)

SUMMARY:
It has been proposed that enriching transfer media with hyaluronan (EmbryoGlue medium) improves pregnancy outcomes compared with media containing lower concentrations of this molecule. However, none of previous studies included preimplantation genetic testing for aneuploidy (PGT-A) embryos. In order to investigate the impact of this hyaluronan-enriched on pregnancy outcomes, it is essential to evaluate its efficacy on euploid-only embryo transfers. The aim of the present study is to evaluate whether a short period of exposure of euploid blastocysts to EmbryoGlue prior to and during transfer positively impact on pregnancy outcomes of frozen embryo transfer (FET) cycles.

DETAILED DESCRIPTION:
The study period will be determined by the completion of the predetermined sample size, with two interim analyses planned when 35% (n=274) and 70% (n=548) of the target sample size is achieved to calculate conditional power. If conditional power is estimated to be lower than 15% at first interim analysis or lower than 30% in the second interim analysis, the trial will be stopped due to futility. The study will be performed in Abu Dhabi-Fertility clinic. During the period of this prospective study, euploid blastocysts of enough quality that have been biopsied only on Day-5 for PGT-A, will be warmed for single blastocyst transfer. The patient´s endometrial preparation protocol for FET will be restricted to HRT only. The study will be double-blinded (blinded to patient and doctor performing transfer).

ELIGIBILITY:
Inclusion Criteria:

* All frozen embryo transfer (FET) cycles with euploid blastocysts biopsied and vitrified on Day 5 after PGT-A.
* Rank of randomization based on embryo quality.
* Only hormonal replacement theraphy (HRT) cycle regimen.
* Women aged 18 years to 46 years.
* Having at least 1 chromosomally normal vitrified blastocyst(s) on Day 5 available for transfer.
* All sperm samples.
* BMI between 18 and 35.

Exclusion Criteria:

* FET cycles with preimplantation genetic testing for monogenic disorders (PGT-M) and for structural rearrangements (PGT-SR).
* FET cycles with mosaic / aneuploid blastocysts.
* FET cycles with unknown outcome.
* FET cycles with Day 6 or Day 7 biopsied blastocysts.
* FET with patients' endometrium preparation with treatments other than HRT.
* FET where PGT-A was performed for gender selection.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 783 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate (LBR) | 41 weeks
  Defined as the delivery if a live infant born after 24 completed weeks of gestation

SECONDARY OUTCOMES:
human chorionic gonadotropin (hCG) positiveness | 10-12 days after embryo transfer
  hCG pregnancy test checks human chorionic gonadotropin (HCG) levels in the blood.
Clinical pregnancy rate | 6 weeks
  ultrasonographic sac visible at 5 gestational weeks
Clinical miscarriage rate | 24 weeks
  spontaneous loss of a clinical pregnancy before 24 weeks of gestation
Ongoing pregnancy rate after 12 weeks | 13 weeks
  viable pregnancy with gestational age more than 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gardner DK, Rodriegez-Martinez H, Lane M. Fetal development after transfer is increased by replacing protein with the glycosaminoglycan hyaluronan for mouse embryo culture and transfer. Hum Reprod. 1999 Oct;14(10):2575-80. doi: 10.1093/humrep/14.10.2575. PMID 10527990
- [Background] Stojkovic M, Kolle S, Peinl S, Stojkovic P, Zakhartchenko V, Thompson JG, Wenigerkind H, Reichenbach HD, Sinowatz F, Wolf E. Effects of high concentrations of hyaluronan in culture medium on development and survival rates of fresh and frozen-thawed bovine embryos produced in vitro. Reproduction. 2002 Jul;124(1):141-53. PMID 12090927
- [Background] Miyano T, Hiro-Oka RE, Kano K, Miyake M, Kusunoki H, Kato S. Effects of hyaluronic acid on the development of 1- and 2-cell porcine embryos to the blastocyst stage in vitro. Theriogenology. 1994;41(6):1299-305. doi: 10.1016/0093-691x(94)90488-5. PMID 16727484
- [Background] Schoolcraft W, Lane M, Stevens J, Gardner D. Increased hyaluronannan concentration in the embryo transfer medium results in a signifcant increase in human embryo implantation rate. In American Society for Reproductive Medicine. 2002 Fertility and Sterility
- [Background] Atkinson B, Woodland E. Embryo Glue: The Use of Hyaluronan in Embryo Transfer Media. Semin Reprod Med. 2021 Mar;39(1-02):24-26. doi: 10.1055/s-0041-1730415. Epub 2021 May 25. PMID 34034352
- [Background] Valojerdi MR, Karimian L, Yazdi PE, Gilani MA, Madani T, Baghestani AR. Efficacy of a human embryo transfer medium: a prospective, randomized clinical trial study. J Assist Reprod Genet. 2006 May;23(5):207-12. doi: 10.1007/s10815-006-9031-7. Epub 2006 Jun 20. PMID 16786421
- [Background] Urman B, Yakin K, Ata B, Isiklar A, Balaban B. Effect of hyaluronan-enriched transfer medium on implantation and pregnancy rates after day 3 and day 5 embryo transfers: a prospective randomized study. Fertil Steril. 2008 Sep;90(3):604-12. doi: 10.1016/j.fertnstert.2007.07.1294. Epub 2007 Oct 23. PMID 17936283
- [Background] Hazlett WD, Meyer LR, Nasta TE, Mangan PA, Karande VC. Impact of EmbryoGlue as the embryo transfer medium. Fertil Steril. 2008 Jul;90(1):214-6. doi: 10.1016/j.fertnstert.2007.05.063. Epub 2007 Sep 4. PMID 17765233
- [Background] Safari S, Razi MH, Safari S, Razi Y. Routine use of EmbryoGlue((R)) as embryo transfer medium does not improve the ART outcomes. Arch Gynecol Obstet. 2015 Feb;291(2):433-7. doi: 10.1007/s00404-014-3416-0. Epub 2014 Aug 24. PMID 25151028
- [Background] Heymann D, Vidal L, Or Y, Shoham Z. Hyaluronic acid in embryo transfer media for assisted reproductive technologies. Cochrane Database Syst Rev. 2020 Sep 2;9(9):CD007421. doi: 10.1002/14651858.CD007421.pub4. PMID 32876946
- [Background] Child et al. A rCT assessing effectiveness of embryoglue in IVF transfer cycles. ASRM abstract 2021.
- [Background] Adeniyi T, Horne G, Ruane PT, Brison DR, Roberts SA. Clinical efficacy of hyaluronate-containing embryo transfer medium in IVF/ICSI treatment cycles: a cohort study. Hum Reprod Open. 2021 Mar 3;2021(1):hoab004. doi: 10.1093/hropen/hoab004. eCollection 2021. PMID 33718621
- [Background] Good practice for recommendation for add-ons in reproductive medicine. ESHRE-working group, 2023.
- [Background] Oron G, Son WY, Buckett W, Tulandi T, Holzer H. The association between embryo quality and perinatal outcome of singletons born after single embryo transfers: a pilot study. Hum Reprod. 2014 Jul;29(7):1444-51. doi: 10.1093/humrep/deu079. Epub 2014 May 8. PMID 24812313
- [Background] Vinals Gonzalez X, Odia R, Naja R, Serhal P, Saab W, Seshadri S, Ben-Nagi J. Euploid blastocysts implant irrespective of their morphology after NGS-(PGT-A) testing in advanced maternal age patients. J Assist Reprod Genet. 2019 Aug;36(8):1623-1629. doi: 10.1007/s10815-019-01496-9. Epub 2019 Jun 4. PMID 31165389
- [Background] Capalbo A, Rienzi L, Cimadomo D, Maggiulli R, Elliott T, Wright G, Nagy ZP, Ubaldi FM. Correlation between standard blastocyst morphology, euploidy and implantation: an observational study in two centers involving 956 screened blastocysts. Hum Reprod. 2014 Jun;29(6):1173-81. doi: 10.1093/humrep/deu033. Epub 2014 Feb 26. PMID 24578475
- [Background] Irani M, Reichman D, Robles A, Melnick A, Davis O, Zaninovic N, Xu K, Rosenwaks Z. Morphologic grading of euploid blastocysts influences implantation and ongoing pregnancy rates. Fertil Steril. 2017 Mar;107(3):664-670. doi: 10.1016/j.fertnstert.2016.11.012. Epub 2017 Jan 6. PMID 28069172
- [Background] Li N, Guan Y, Ren B, Zhang Y, Du Y, Kong H, Zhang Y, Lou H. Effect of Blastocyst Morphology and Developmental Rate on Euploidy and Live Birth Rates in Preimplantation Genetic Testing for Aneuploidy Cycles With Single-Embryo Transfer. Front Endocrinol (Lausanne). 2022 Apr 13;13:858042. doi: 10.3389/fendo.2022.858042. eCollection 2022. PMID 35498424
- [Background] Xiao Y, Wang X, Gui T, Tao T, Xiong W. Transfer of a poor-quality along with a good-quality embryo on in vitro fertilization/intracytoplasmic sperm injection-embryo transfer clinical outcomes: a systematic review and meta-analysis. Fertil Steril. 2022 Dec;118(6):1066-1079. doi: 10.1016/j.fertnstert.2022.08.848. Epub 2022 Oct 14. PMID 36244848
- [Background] Brosens JJ, Salker MS, Teklenburg G, Nautiyal J, Salter S, Lucas ES, Steel JH, Christian M, Chan YW, Boomsma CM, Moore JD, Hartshorne GM, Sucurovic S, Mulac-Jericevic B, Heijnen CJ, Quenby S, Koerkamp MJ, Holstege FC, Shmygol A, Macklon NS. Uterine selection of human embryos at implantation. Sci Rep. 2014 Feb 6;4:3894. doi: 10.1038/srep03894. PMID 24503642
- [Background] C. Jennison and B. W. Turnbull, "Group Sequential Methods with Applications to Clinical Trials," Chapman & Hall/CRC, Boca Raton, 2000.